#### INFORMED CONSENT/ASSENT FORM

Consent form version date: September 6, 2022

# Girls Invest: A Mobile-Enabled Economic Empowerment Intervention for Girls Quantitative Surveys

This study is being conducted primarily by investigators at San Diego State University (Dr. Elizabeth Reed).

The study is sponsored by the National Institutes of Health.

#### **IMPORTANT THINGS TO KNOW ABOUT THIS STUDY:**

We are inviting you to join this research study. The purpose of this research is to see whether *Girls Invest* provides girls with support to reach their future goals. *Girls Invest* aims to support girls' health knowledge, improve career and educational expectations, increase girls' knowledge about finances, and increase girls' safety in relationships to make sure girls have healthy intimate relationships where they are supported to reach their future goals. The program addresses many things related to girls' family life, friends, choices about money, school, education, training, employment, relationships, and future goals. *Girls Invest* provides information through an app over a mobile phone or tablet. As part of the program, girls are also enrolled into a savings account and receive funds deposited into the account based on their completion of the different training levels in the app.

If you agree to join the study, we will ask you to a) complete two surveys, one today and one in 6 months, b) download an app and complete training modules on various topics (as described in more detail below), c) open a savings account, and d) recruit at least one friend to participant in the study with you. Participation in the surveys will take approximately 45 minutes. Time to complete the training modules in the app will vary (approximately 40 minutes for each of five levels of training) and will depend on your previous knowledge of a topic area. Participants receive \$10 to open a savings account and \$20 deposited into their savings account after the completion of each level of training. For completing the study surveys, you will also receive a reimbursement for your time (\$25 for the first survey and \$30 for the second survey). Participants who recruit a friend (index participants) will receive a \$25 gift card upon successful enrollment of a friend; the gift card will be provided when the friend has completed the baseline survey and the savings account application.

You do not have to join this study to answer our questions, but if you do, you will be helping us better understand whether *Girls Invest* is a program that supports girls' future goals and expectations, especially in increasing girls' access to opportunities for education/training, career, and financial well-being, while also reducing their risk for poor health. Participants may benefit from obtaining more information about relationships, information on health issues important to girls, and how to save and invest money, including how to apply for educational loans and scholarships, how to lease a car, and how to rent an apartment. Participants may also benefit from getting a savings account with money deposited.

One reason you may decide to join the study may be to gain access to this information or to set up a savings account. You may also decide you are not interested to join the study because you will be asked personal questions (sometimes sensitive questions about sex, relationships etc.) as part of a questionnaire that you need to complete twice during your participation in the study. However, the information you provide will be confidential and only linked to your study ID (See more details on this below in the section called: "Will my information be private?).

#### INFORMED CONSENT/ASSENT FORM

Consent form version date: September 6, 2022

We will give you more details about why we are doing this study, what we will ask you to do, the possible risks and benefits of allowing us to ask you questions. We will explain the other choices you have. We will also give you any other information that you need to make an informed choice about joining this study.

The following information is a more complete description of the study. Please read this description carefully. We want you to ask us any questions that will help you decide whether you want to join this study. If you join the study, we will give you a signed copy of this form to keep so that you have information for later if you need it.

#### WHO SHOULD I CONTACT IF I HAVE QUESTIONS OR CONCERNS?

Principal Investigator: Dr. Elizabeth Reed

Department: Health Promotion and Behavioral Sciences

Address: School of Public Health, San Diego State University. 5500 Campanile Drive San Diego, CA 92182

Email: ereed@sdsu.edu

#### WE ARE INVITING YOU TO JOIN THIS RESEARCH STUDY.

We are inviting you because you are participating in one of our collaborating schools or community programs. You may have also indicated that you are between 15-22 years old, are female, live in either City Heights, San Ysidro, Southeast San Diego, El Cajon, Vista, Escondido, Murietta, Chula Vista, National City (or another neighborhood in the San Diego County region), have a smartphone with internet access, and are willing to open a savings account.

Up to 240 participants will be included as part of this study.

Research is not the same as treatment, or other medical or psychological care or therapy. The purpose of research is to answer scientific questions.

You do not have to be in this study. You are free to say "yes" or "no", or to drop out of the study after joining.

If you heard about the study or were referred to the study while receiving clinical care, please note that this research study is not related to your clinical care. Your participation (or decision not to participate) will not affect your clinical care. If you consent to participate in the study, but then later, you decide to end your participation in the study, this will also not affect your clinical care.

#### WHY ARE WE DOING THIS STUDY?

The purpose of this research is to figure out how to better meet the needs of teen girls. We would like girls to take part in the *Girls Invest* program so that we can see whether it is beneficial to support girls. *Girls Invest* aims to support girls' knowledge of their health, improve career expectations, increase girls' knowledge about finances, and to increase girls' safety in relationships to ensure girls have healthy intimate relationships, given that having healthy relationships is important for girls to be able to invest in their future goals. Through an app on a smartphone, *Girls Invest* addresses many aspects of girls' family life, friends, choices about money, school, education, training, employment, relationships, and future goals. As we mentioned before, the program also enrolls girls into a savings account and provides deposits into the account based on their completion of the app-based program, which is meant to be fun and interactive.

#### WHAT IS THE TIME COMMITMENT IF I JOIN THIS RESEARCH STUDY?

#### INFORMED CONSENT/ASSENT FORM

Consent form version date: September 6, 2022

Your participation will last about 45 minutes during completion of each survey. Time to complete the app-based training modules will vary based on the individual but will be approximately 40 minutes per training level for each of 5 trainings (3-4 hours total). Once you take each training, you will have access to the information at any time and can go back to any topic area of interest using the menu in the app. This information will be available to you through the app for as long as you have access to the app (even after your participation in the study ends).

The research scientist could take you out of the study at any time. This would happen if:

- They think it is in your best interest to stop being in the study.
- You are not willing or able to do all the things needed in the study.
- The whole study stops.

If you stop participating in this study, information collected before you stopped being in the study will not be included in the analysis of study results. You can contact Dr. Elizabeth Reed (508-212-1517, <a href="mailto:ereed@sdsu.edu">ereed@sdsu.edu</a>) if you wish to withdraw from the study, and you can also request that any data you have provided be withdrawn and destroyed.

#### WHAT WILL I BE ASKED TO DO IN THIS RESEARCH STUDY?

- -You will be asked to download a mobile app and complete an interactive program with five different training modules. The *Girls Invest* app contains information on things related to girls' family life, friends, choices about money, school, education, training, employment, future goals, and relationships, given that having healthy relationships is important for girls to be able to invest in their future goals. Here are the topics covered:
  - 1) How does being a girl affect our health and career/educational choices? This level of training covers health issues like physical activity and body image. It also discusses topics relevant to girls' decisions for their future education and career goals.
  - 2) Money, relationships, and your future what do healthy relationships look like? How might things like money influence relationships?
  - 3) Everything you need to know about applying for future educational loans and scholarships. Many people have heard myths about who is eligible and what is needed. We provide information so you can be an expert.
  - 4) Finance 101: Everything you should know about your money and what to do with it to support your future.
  - 5) Young women working: How to get the job, develop your resume, identify good references, and other things to help girls develop their career goals.

As you advance through five levels, you will be provided with funds deposited into a savings account, totaling \$110. The *Girls Invest* program will be done in stages. You may be asked to participate immediately or you may wait up to 6 months prior to participating in the *Girls Invest* program.

-In order to receive the funds deposited into a savings account from completion of the Girls Invest app training modules, you will need to apply for a savings account with the project-affiliated credit union or bank. You will receive information on how to apply. You can apply online or in-person. You will need a

#### INFORMED CONSENT/ASSENT FORM

Consent form version date: September 6, 2022

photo ID and to provide your study ID to apply. After 6 months of your participation in the study, we will obtain information from the bank on the final amount in your account. After your study participation is over, we will no longer have access to information about your account. However, you will be able to keep this account on your own and keep all of the money deposited as a result of your participation in the *Girls Invest* trainings. You can choose to make additional deposits into the account or to withdraw existing funds at any time.

- -You will complete two confidential surveys on girls' health. We will do one survey now and an additional survey in approximately 6 months. These questionnaires will help us obtain information to understand whether the Girls Invest program has any improvement on girls' expectations and investment for their futures. We will be asking you questions about you (your age, where you live, your education, your household), your knowledge of finance and confidence to manage financial issues on your own, your expectations for future education and career goals, your relationships (including male partners and negative experiences or violence experienced with these partners), sexual and reproductive health behavior, and alcohol/substance use. Some of the questions may be hard to answer. You may refuse to answer any questions. The survey will be taken using the Girls Invest app, which reads the questions to you, and you will respond to the questions on your phone using the app. We will provide you with headphones so you can take the survey privately without others hearing the questions. We encourage you to find a private space (without others around you) to take the survey where you will not be interrupted. We can provide space if you would like. All information you provide to the study will be kept confidential and private. In other words, the information you provide during the survey will not be shared with anyone outside the research team. The information you provide in the survey will be identified with an ID number only and not your name.
- As part of the study, you will be contacted every two months so that we make sure we have updated contact information for you. At this time, we will also check in and see how your participation is going and if you have any questions or need for referrals. We will also ask that you provide 3 alternate contacts, who can be friends or anyone else that you give us permission to contact to be able to reach you in case your phone number changes. We will also contact you to remind you to take the follow-up survey.
- -Based on your participation in this study, there may be a chance that we may ask you about whether you may be interested in also participating in a follow-up interview that will ask about what you like or do not like about the *Girls Invest* program. Interviews will also ask girls how the program influenced them. However, you are not obligated to participate in this follow-up interview as part of this current study.

# WHAT ARE THE RISKS OR DISCOMFORTS INVOLVED IN THE RESEARCH? Risks associated with the study: Loss of Confidentiality

Even though we will take measures keep information collected in the surveys private, there is a possible risk of loss of privacy.

(See "Will my information be private" for more information on how the information collected will be kept confidential).

#### What other risks are associated with this study?

#### INFORMED CONSENT/ASSENT FORM

Consent form version date: September 6, 2022

Because of the personal nature of the questions to be asked, you might reflect on unpleasant memories while participating in an interview. For example, you may feel uncomfortable answering questions about your personal attitudes, beliefs and behaviors, including financial information or sexual behaviors. Some issues may be uncomfortable and could have an emotional impact; however, you may decline to answer any question you do not wish to answer. If after participating, and you would like to talk to someone, we will arrange that for you. Remember, however, that all of the information that you provide is confidential. None of the study's reports or publications will use your name or any other identifying information. Only authorized members of the research team will have access to your information that could identify you as a participant in this research.

As part of participating in *Girls Invest*, you will receive a savings account with funds deposited into it as you complete the trainings on the app. There is a risk that if others find out about your account (e.g. you tell them about it, or you use the money you earned in some way so that they find out), they may ask you about how you have it or pressure you to give money to them. Given that the app is on your phone, others may see that you have this app; however, because the app has a password only you will be able to log onto the app. The information you provide via the surveys you take over the app will not be able to be accessed after you submit each response. We encourage you to take these surveys in a private location, however, and we can provide you with a private location that is convenient for you if you need one.

Dr. Reed (the lead researcher from the San Diego State University which is overseeing this study) has a **Certificate of Confidentiality** from the Federal government that will help us protect the privacy of research subjects enrolled in this study. The Certificate of Confidentiality allows the investigator and others who have access to research records to refuse to disclose identifying information on research participants in any civil, criminal, administrative, legislative, or other proceeding, whether at the federal, state, or local level.

A Confidentiality Certificate does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If you have given your consent for an insurer or employer to obtain information about you, the investigator may not use the Certificate of Confidentiality to withhold this information. A Certificate of Confidentiality also does not prevent an investigator from disclosing information about you to prevent serious harm to yourself or others, such as reporting to the authorities incidents of child abuse or elder abuse.

You will be able to call the San Diego State University Institutional Review Board office (contact information is below) to discuss any discomfort that you experienced during your study participation.

Because this is a research study, there may also be some unknown risks that are currently unforeseeable. You will be informed of any significant new findings.

#### **ARE THERE ANY BENEFITS TO PARTICIPATION?**

You may benefit from obtaining the information in the app, such as information about financial matters, ways to achieve career and educational goals, increased knowledge about sexual and reproductive health and knowledge of healthy versus unhealthy relationship behaviors. You may also benefit from starting a savings account and having money deposited into that account that you can use or invest.

While you will access information and get a savings account with money deposited to your account, we do not know for sure if or how you will benefit from these things. By joining this research study, you are helping us to find out whether *Girls Invest* may benefit girls your age. Your participation will also be used to help us improve *Girls Invest*.

#### INFORMED CONSENT/ASSENT FORM

Consent form version date: September 6, 2022

Otherwise, there are no direct and immediate benefits from participation in this study, other than any satisfaction that you may gain from the opportunity to contribute to research that aims to improve girls' health and well-being. More generally, it is our hope that the knowledge we gain from you and other participants will help us develop better health interventions among youth.

#### ARE THERE ANY ALTERNATIVES TO JOINING THIS RESEARCH STUDY?

An alternative is to not join the research study.

#### WILL MY INFORMATION BE PRIVATE?

<u>Girls Invest program</u>: The app will require a username and log-in which will contain only your unique identifier (an ID that we provide to you that will be used to identify you instead of your name). The information you provide via the surveys you take over the app will not be able to be accessed after you submit your responses. We encourage you to take these surveys in a private location, however, and we can provide you with a private location that is convenient for you if you need one. Your information collected as part of this research will not be used or distributed for future research studies without first contacting you to obtain your consent.

<u>Surveys</u>. Your individual participant survey data will be obtained from structured 45-minute surveys by a self-administered program in the app. Trained research assistants will provide any needed technical assistance for the completion of the surveys through the app. If needed, research staff can assist by setting up a meeting with you to help you complete the survey over the app. All survey data will be uploaded and connected to participants by study ID only. In other words, only your ID (not your name) will be associated with the data you provide through the survey. We will have a separate sheet that we will keep in a locked file that has all participant names and associated study ID, which will only be used for when we need to contact you, like to remind you to take the follow-up survey.

Research records will be stored in a locked electronic file and will only be accessible to research staff. Research records with identifying information will be destroyed three years after the end of this study. Research records may be viewed by the San Diego State University Institutional Review Boards as well as other authorities if any events are reported where you report being harmed by study participation or if you report serious harm to yourself or others, such as reporting to the authorities incidents of child abuse or elder abuse. Under law, we must report information about known or reasonably suspected incidents of abuse or neglect of a child, dependent adult or elder, including physical, sexual, emotional, and financial abuse or neglect. If any investigator has or is given such information, he or she may be required to report such information to the appropriate authorities. If you report at any time during study participation of your intent to harm yourself or someone else, we are mandated by law to report this intent. If you report intentions to harm yourself, we will be required to ensure that you receive attention and treatment by immediately taking you to appropriate services.

#### DO I HAVE TO JOIN THIS STUDY?

You do not have to join this research study. If you choose not to participate, there is no penalty or loss of benefits to which you are otherwise entitled. If you heard about this study at school or in a class of yours, participation in the study has no effect on your class grades. Additionally, you may choose to stop participating at any time without penalty or loss of benefits to which you are otherwise entitled. If you would like to withdraw your participation, you can do so by informing any of the project staff in person or contacting Dr. Reed (508-212-1517, ereed@sdsu.edu).

#### INFORMED CONSENT/ASSENT FORM

Consent form version date: September 6, 2022

You will be told if any important new information is found during the course of this study that may affect you wanting to continue.

#### WILL I BE TOLD ABOUT THE RESEARCH RESULTS?

We will not contact you with results of this study after this study is completed. The findings of this study will be used to improve the *Girls Invest* program and prepare to provide the program to a larger population of girls in the future.

#### WILL IT COST ME ANYTHING IF I JOIN THE RESEARCH?

There are no costs to you to participate in the study.

#### WILL I BE PAID IF I JOIN THE RESEARCH?

In compensation for your time and travel expenses, you will receive a \$25 Amazon e-gift card for completing the first survey and an additional \$30 Amazon e-gift card at follow-up upon completion of the follow-up survey.

Additionally, up to \$110 will be deposited into a savings account in increments. The total amount of money deposited will depend on how many training modules you complete in the mobile app.

#### ANY APPARENT OR POTENTIAL CONFLICT OF INTEREST

We are not aware of any information that may cause the researchers to do their work in a way that will interfere with the study conduct and findings.

#### WHOM DO I CONTACT IF I HAVE QUESTIONS OR CONCERNS?

If you have other questions or research-related problems, you may reach Dr. Reed at 508-212-1517 or ereed@sdsu.edu. You may call the SDSU Institutional Review Board Office at (619) 594-6622 to inquire about your rights as a research subject or to report research-related problems.

At any time during the research, you can contact the IRB for questions about research rights, to discuss problems, concerns, give suggestions, or to offer input.

#### **CONSENT/ASSENT TO PARTICIPATE**:

This research has been approved by the San Diego State University Institutional Review Board, as signified by the Board's stamp. The IRB must review the consent form yearly. The IRB approval expires on the date indicated by the stamp in the upper right-hand corner of this document.

Your signature below indicates that you have read the information in this document and have had a chance to ask any questions you have about the study. Your signature also indicates that you agree to join the study and that the study team has told you that you can change your mind and withdraw your consent to participate at any time. The investigator or a member of his/her research team has provided you with a copy of this consent form with information about who to contact in the event you have questions.

### **INFORMED CONSENT/ASSENT FORM**

Consent form version date: September 6, 2022

| Check here is <u>assent</u> is being provided (participant is under 18 years of age): | |
|---|---|
| Name of Participant (please print) | |
| Signature of Participant | Date |
| Signature of Investigator | Date |